CLINICAL TRIAL: NCT00816673
Title: Phase II Study of Sleep Inducing And Maintaining Efficacy Of Circadin In Elderly Insomniacs.
Brief Title: Sleep Inducing And Maintaining Efficacy Of Circadin In Elderly Insomniacs
Acronym: Neu I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Tali Nir Director Clinical and Regulatory Affairs, Neurim Pharmaceuticals Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neurim I
Record Dates: First submitted 2008-12-31; First posted 2009-01-05 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Primary Insomnia
Keywords: Insomnia; Primary insomnia; sleep latency; non restorative sleep; sleep quality; Double-Blind; Placebo Controlled; Parallel-Group; Sleep Laboratory Study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo Circadin
- Circadin (Experimental)
  Interventions: Drug: Circadin

INTERVENTIONS:
Drug: placebo Circadin — Placebo tabs of Prolonged release melatonin
  Arms: placebo
Drug: Circadin — prolonged release melatonin 2 mg taken daily 2 hours before bed-time for 3 weeks
  Other Names: ATC code: N05CH01
  Arms: Circadin

SUMMARY:
The aim of this placebo controlled study is to investigate the effect of 2 mg melatonin Slow Release (Circadin®) on the sleep/wake cycle in elderly insomniac out-subjects, aged 55 years or more.

DETAILED DESCRIPTION:
Circadin® is a newly developed slow release galenic formulation of melatonin, producing overall levels of melatonin comparable to those observed in a control population, when administered to patients with deficiency in melatonin; thus it deserves more clinical and paraclinical investigations for establishing efficacy in inducing and maintaining sleep and for safety. Since, on the one hand, the endogenous substance melatonin has beneficial effects on sleep in man and, on the other hand, there is a decrease in melatonin secretion in elderly people, substitution therapy in elderly insomniacs would be a desirable therapy.

The aim of this placebo controlled study was to investigate the effect of 2 mg Melatonin Slow Release (Circadin®) on the sleep/wake cycle in elderly insomniac out-subjects, aged 55 years or more. Sleep was assessed by means of polysomnography (hypnographic results), all-night sleep EEG spectral analysis (functional and quantitative results of sleep EEG), actimetry (SomnitorTM), wake EEG and sleep/wake quality questionnaires. Vigilance and cognitive skills were assessed by means of psychomotor and neurocognitive tests derived from the Leeds psychomotor test battery (vigilance and arousal) and TEA battery (attention).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female, aged ≥ 55 years, suffering from primary insomnia according to DSM-IV criteria (307.42)

Exclusion Criteria:

* According to DSM-IV, subjects belonging to the following groups are excluded: 780.59; 307.45; 307.47; 780.xx (Appendix 2);
* Use of benzodiazepines or other hypnotics during the preceding 1 month with a frequency of more than 2 times a week and lasting more than 2 weeks;
* Severe neurological, psychiatric or sleep disorders;
* Other serious diseases;
* Taking more than 1/2 l of alcohol, more than 3 cups of coffee or more than 10 cigarettes per day .
* Subjects who need beta blockers as a treatment.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1996-09; Primary Completion 1997-05 (Actual); Study Completion 1997-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul MACHER, MD, Principal Investigator — Forenap
Locations (1):
- FORENAP, Centre Hospitalier de Rouffach, France